CLINICAL TRIAL: NCT03745417
Title: Efficacy and Safety of Expanded Umbilical Cord Mesenchymal Stem Cells On Patients With Moderate to Severe Psoriasis
Brief Title: Efficacy and Safety of Expanded UCMSCs On Patients With Moderate to Severe Psoriasis
Acronym: UCMSCs
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Chuanjian Lu, Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2018-11
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Mesenchymal Stromal Cells; Psoriasis; Drug Effect; Drug Toxicity
Keywords: Psoriasis; Umbilical cord Mesenchymal Stem Cells
MeSH Terms: conditions — Psoriasis; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCMSCs group (Experimental): Umbilical cord mesenchymal stem cells intravenous injection at a dose of 2 million cells/kg at week 0,week 2,week 4,week 6,week 8 with a duration for treatment for 12 weeks.
  Interventions: Biological: Umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Umbilical cord mesenchymal stem cells — Umbilical cord mesenchymal stem cells were infused intravenously at a dose of 2 million cells/kg.
  Other Names: UCMSCs

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Expanded Umbilical Cord Mesenchymal Stem Cells on patients with moderate to severe psoriasis. Any adverse events related to UCMSCs infusion will be monitored.The primary outcome is the improvement rate of PASI(Psoriasis Area and Severity Index) and treatment response will be computed from PASI before and after UCMSCs infusion.

DETAILED DESCRIPTION:
Psoriasis is an immune-mediated, genetic disease manifesting in the skin or joints or both. Numerous topical and systemic therapies are available for the treatment of psoriasis. Treatment modalities are chosen on the basis of disease severity, relevant comorbidities, patient preference. For moderate to severe psoriasis, phototherapy, systemic therapy and biologic immune modifying agents are recommended, but all of them have some drawbacks or limitations. Until now, no curative treatment is available. Therefore, it is important to find new treatment for psoriasis. Mesenchymal stem cells (MSCs) are a kind of adult stem cells that can differentiate into bone, cartilage and adipose cells. Umbilical cord Mesenchymal Stem Cells were isolated from umbilical cord matrix and were reported to treat moderate to severe psoriasis vulgaris and psoriasis arthritis successfully by case reports. For the mechanism of the disease, involvement of the immune system in psoriasis is now widely accepted. Mesenchymal stem cells (MSCs) are found to have the function of immunomodulation, migration to skin lesions, limitation of autoimmunity. Therefore, investigators supposed that the injection of UCMSCs could be beneficial for treatment of moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1．moderate to severe psoriasis vulgaris ( PASI > 7 or BSA >10% ) 2．18 to 65 years old 3．written/signed informed consent

Exclusion Criteria:

1. guttate psoriasis, inverse psoriasis or exclusively associated with the face
2. Acute progressive psoriasis, and erythroderma tendency
3. current (or within 1 year) pregnancy or lactation
4. current significant anxiety or depression with the Self-rating Anxiety Scale (SAS) > 50 or the Self-rating Depression Scale (SDS) > 53, or with other psychiatric disorders
5. With history of primary cardiovascular, respiratory, digestive, urinary, endocrinologic and hematologic diseases, which can't be controlled through ordinary treatments. Those who with malignant diseases, infections, electrolyte imbalance, acid-base disturbance. Patients with clinical test results listed below: abnormal serum calcium level ( Ca2+ > 2.9 mmol/L or < 2 mmol/L);AST or ALT 2 times more than normal upper limit; Creatinine and cystatin C more than normal upper limit; Hemoglobin elevates 20g/L more than normal upper limit,or hemoglobin reduction to anemia; Platelet count less than 75.0*10^9/L; White blood cell less than 3.0*10^9/L; Or any other abnormal laboratory test results, assessed by investigators, that are not suitable for this clinical study
6. Patients with malignant tumors, or when they were enrolled with abnormal tumor markers or with other organ dysfunction
7. allergy to anything else ever before;
8. current registration in other clinical trials or participation within a month;
9. topical treatments (i.e. corticosteroids or retinoic acid or Vitamin D analogs ) within 2 weeks; systemic therapy or phototherapy (ultraviolet radiation B,UVB) and psoralen combined with ultraviolet A (PUVA) within 4 weeks; biological therapy within 12 weeks;
10. medical conditions assessed by investigators, that are not suitable for this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-08-31 (Estimated); Primary Completion 2022-08-28 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
PASI score improvement rate | 12 weeks (plus or minus 3 days) after treatment
  PASI score improvement rate = (PASI score before intervention - PASI score after intervention)/PASI score before intervention ×100%

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index(PASI) | 12 weeks (plus or minus 3 days) after treatment
  The improvement in PASI score from baseline after treatment. PASI scores the average redness, thickness, and scaliness of the lesions (0-4 scale), weighted by the area of involvement. PASI scores range from 0 to 72.
Relapse rate in treatment period / follow-up period | During the treatment period of 12 weeks / follow-up period of 12 weeks after treatment period
  Relapse can be defined only for patients who achieve PASI50，and occurs when the improvement in the PASI score falls below 50% from the baseline PASI score.
PASI-50 | 12 weeks (plus or minus 3 days) after treatment
  The proportion of patients who achieve at least 50% improvement in PASI score from baseline. PASI scores the average redness, thickness, and scaliness of the lesions (0-4 scale), weighted by the area of involvement. PASI scores range from 0 to 72.
PASI-75 | 12 weeks (plus or minus 3 days) after treatment
  The proportion of patients who achieve at least 75% improvement in PASI score from baseline. PASI scores the average redness, thickness, and scaliness of the lesions (0-4 scale), weighted by the area of involvement. PASI scores range from 0 to 72.
Pruritus Scores on the Visual Analogue Scale | 12 weeks (plus or minus 3 days) after treatment
  Pruritus Scores on the Visual Analogue Scale
the Body Surface Area (BSA%) | 12 weeks (plus or minus 3 days) after treatment
  the Body Surface Area
the Dermatology Life Quality Index（DLQI） | 12 weeks (plus or minus 3 days) after treatment
  the score of Dermatology Life Quality Index. Dermatology Life Quality Index (DLQI) is a self-administered 10-item questionnaire. It covers Symptoms and feelings, Daily activities, Leisure, Work and school, Personal relationships, and Treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China